CLINICAL TRIAL: NCT01112072
Title: Randomized Study of Safety and Effectiveness of Corneal Collagen Crosslinking and Intacs for Treatment of Keratoconus and Corneal Ectasia
Brief Title: Corneal Collagen Crosslinking and Intacs for Keratoconus and Ectasia
Acronym: CXL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEI-Intacs-CXL
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: keratoconus; corneal ectasia; collagen crosslinking; riboflavin; cornea; ultraviolet
MeSH Terms: conditions — Keratoconus; Corneal Diseases | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intacs combined with CXL (Active Comparator): Intacs placement followed by collagen crosslinking with UV light and riboflavin
  Interventions: Drug: Riboflavin
- Intacs followed by CXL (Active Comparator): Intacs placement, to be followed by corneal collagen crosslinking with UV light and riboflavin 3 months later
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Corneal epithelium removed followed by riboflavin drop administration every 2 minutes for 30 minutes followed by UV light exposure with additional riboflavin administration every 2 minutes for 30 minutes. Subjects will be randomized to receive Intacs placement either immediately before CXL or 3 months before CXL.
  Other Names: Intracorneal Ring Segments; Cornea Collagen Crosslinking

SUMMARY:
This study will determine the efficacy of corneal collagen crosslinking (CXL) combined with Intacs for the treatment of keratoconus and corneal ectasia. The goal of CXL is to decrease the progression of keratoconus, while Intacs has been shown to decrease corneal steepness in keratoconus. This study will attempt to determine the relative efficacy of the two procedures either performed at the same session versus CXL performed 3 months after Intacs.

DETAILED DESCRIPTION:
The purpose of this is to ascertain the possible additive effect of the two treatments to both improve the quality of the corneal optics (i.e. improve corneal topography regularity) and to stabilize the cornea. Previous investigations have shown that Intacs surgery, indeed, does improve corneal topography and improve contact lens tolerance and spectacle corrected visual acuity, as well as uncorrected visual acuity in some patients. Investigations of CXL have shown the procedure not only to decrease keratoconus progression, but also to decrease the steepness of the cone and improve uncorrected and best corrected visual acuity in some cases. Since the mechanism of improvement differs between the procedures, this suggests a potential additive effect of the two on the patient's ultimate visual outcome. Thus, the patient would be afforded two potential benefits: (1) the potential of a more robust visual outcome and (2) stabilization of the keratoconic cornea on the longer term.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Having a diagnosis of keratoconus or corneal ectasia after corneal refractive surgery (e.g., LASIK, photorefractive keratectomy [PRK], or epi-LASIK)
* Subjects who meet the manufacturer's nomogram recommendations for Intacs segments
* Topography consistent with keratoconus or post-surgical corneal ectasia.
* BSCVA worse than 20/20 (<55 letters on ETDRS chart)

Exclusion Criteria:

* Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme.
* Corneal pachymetry ≤ 400 microns at the thinnest point measured by Pentacam in the eye(s) to be treated when the isotonic riboflavin solution is used or ≤ 300 microns when the hypotonic riboflavin us used, provided that the corneal thickness after treatment with the hypotonic riboflavin solution is > 400 microns. Corneal pachymetry ≤ 450 microns at the proposed insertion site for the Intacs
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications
* History of corneal disease
* History of chemical injury or delayed epithelial healing in the eye(s) to be treated.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Subjects with nystagmus or any other condition that would prevent a steady gaze during the CXL and Intacs treatment or other diagnostic tests.
* Subjects with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-04; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum keratometry | 1 year

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, M.D., Principal Investigator — Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institute, Teaneck, New Jersey, United States